CLINICAL TRIAL: NCT02938377
Title: Alcohol Research Consortium in HIV-Intervention Research Arm
Acronym: ARCH-IRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Karen Cropsey, Principal Investigator, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F160706007
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: HIV Positive; Alcohol Use
MeSH Terms: conditions — HIV Seropositivity; Alcohol Drinking | interventions — Cognitive Behavioral Therapy; Counseling; Ethanol; APT

STUDY DESIGN:
Intervention Model Description: Participants were given varying levels of treatment depending on their alcohol use.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- No dx of alcohol use disorder, panic or depression (Active Comparator): Computerized Brief Intervention (CBI)- a video about alcohol abuse
  Interventions: Behavioral: Computerized Brief Intervention (CBI)
- Risky drinking, no dx of AUD, has panic or depression (Active Comparator): Computerized Brief Intervention (CBI)- a video about alcohol abuse, plus 4 sessions of counseling called Motivational Enhancement Therapy
  Interventions: Behavioral: Computerized Brief Intervention (CBI); Behavioral: CBT4CBT
- Dx of AUD with or without panic or depression (Active Comparator): Computerized Brief Intervention (CBI)- a video about alcohol abuse, plus 4 sessions of counseling called Motivational Enhancement Therapy plus a recommendation for Alcohol Pharmacotherapy (APT). The drugs recommended in the APT are all standard of care drugs for alcohol treatment and are not under study in this protocol.
  Interventions: Behavioral: Computerized Brief Intervention (CBI); Behavioral: CBT4CBT; Drug: Recommendation and Counseling for Alcohol Pharmacotherapy

INTERVENTIONS:
Behavioral: Computerized Brief Intervention (CBI) — A video which emphasizes personal responsibility for change, uses empathy as a counseling style, and enhances self-efficacy. Depending on alcohol dependence level, four different CBI versions may be shown over two visits.
  Other Names: CBI
Behavioral: CBT4CBT — 9 computerized modules delivered at the participant's pace
  Other Names: Cognitive Behavioral Therapy
  Arms: Dx of AUD with or without panic or depression; Risky drinking, no dx of AUD, has panic or depression
Drug: Recommendation and Counseling for Alcohol Pharmacotherapy — The APT algorithm will utilize the four FDA approved APTs for the treatment of alcohol use disorder. The treatment of the patient is part of routine care.
  Other Names: Recommendation for APT
  Arms: Dx of AUD with or without panic or depression

SUMMARY:
Aim 1: Examine effects of algorithm-guided alcohol treatment on alcohol consumption and alcohol use Disorders (AUD) symptoms.

Aim 2: Examine effects of algorithm-guided alcohol treatment on retention in HIV care and HIV-related outcomes.

Aim 3: Examine effects of algorithm-guided alcohol treatment on comorbid conditions

DETAILED DESCRIPTION:
Aim 1: Examine effects of algorithm-guided alcohol treatment on alcohol consumption and alcohol use Disorders (AUD) symptoms. Hypothesis 1A: Patients who are treated using algorithm-guided alcohol treatment will decrease drinking quantity and or frequency compared to pre-algorithm levels. Hypothesis 1B. Patients who are treated using algorithm-guided treatment will decrease current AUD symptoms compared to pre-algorithm symptoms levels.

Aim 2: Examine effects of algorithm-guided alcohol treatment on retention in HIV care and HIV-related outcomes. Hypothesis 2A. Patients treated using algorithm-guided treatment will increase adherence to clinic visits and HIV medications compared to pre-algorithm levels. Hypothesis 2B. Patients who receive algorithm-guided treatment will have improved HIV biomarkers (e.g., CD4 and VL). Hypothesis 3B. There will be a positive relationship between VL and alcohol consumption measured by self-report and PEth level.

Aim 3: Examine effects of algorithm-guided alcohol treatment on comorbid conditions (e.g., depression, anxiety, HCV, other drug use disorders). Hypothesis 3A: Persons living with HIV (PLWH) with co-morbid depression and anxiety receiving algorithm-guided treatment will have better alcohol, mental health and HIV treatment outcomes compared to similar individuals in SC. Hypothesis 3B: PLWH with comorbid HCV receiving algorithm-guided treatment will have improved FIB4 results and reduced likelihood of HCV recurrence compared to persons in SC. Hypothesis 3C: Other drug use will decrease among those receiving algorithm-guided treatment vs SC.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years or older;
* Receiving HIV care at the UAB, UW or UCSD clinics and not anticipating changing clinics over the next 12 months;
* AUDIT-C score > 3 women or > 4 men at time of PRO.

Exclusion Criteria:

* Non-English speaking;
* Acutely suicidal, manic, acutely intoxicated, or otherwise not stable enough to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4985 (Actual)
Dates: Start 2017-11-06 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2023-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Harborview Medical Center; 2 West Clinic; UW Center for AIDS, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- No dx of Alcohol Use Disorder, Panic or Depression: This arm received standard of care services at each clinic.
Period: Overall Study
Arm/Group | Risky Drinking, no dx of AUD, Has Panic or Depression | Dx of AUD With or Without Panic or Depression | No dx of Alcohol Use Disorder, Panic or Depression
Started | 115 | 27 | 4843
Completed | 115 | 27 | 4843
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- No dx of Alcohol Use Disorder, Panic or Depression: This arm will receive standard of care services at each clinic.
- Total: Total of all reporting groups
Arm/Group | Risky Drinking, no dx of AUD, Has Panic or Depression | Dx of AUD With or Without Panic or Depression | No dx of Alcohol Use Disorder, Panic or Depression | Total
Number analyzed (Participants) | 115 | 27 | 4843 | 4985
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12) | 45 (11) | 49 (12) | 47 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 3 | 969 | 994
  Male | 93 | 24 | 3874 | 3991
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 45 | 9 | 1839 | 1893
  Non-Hispanic Black | 55 | 8 | 2151 | 2214
  Hispanic | 11 | 9 | 649 | 669
  Other | 4 | 1 | 204 | 209

OUTCOME MEASURES:

1. Primary Outcome: Audit-C Score on a Scale
Description: Difference in Audit-C score, pre and post intervention. The AUDIT-C is scored on a scale of 0-12 (scores of 0 reflect no alcohol use). In men, a score of 4 or more is considered positive; in women, a score of 3 or more is considered positive. Generally, the higher the AUDIT-C score, the more likely it is that the patient's drinking is affecting his/her health and safety.
Time Frame: 18 month window
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Dx of AUD With or Without Panic or Depression: Computerized Brief Intervention (CBI)- a video about alcohol abuse, plus 4 sessions of counseling called Motivational Enhancement Therapy plus a recommendation for Alcohol Pharmacotherapy (APT). The drugs recommended in the APT are all standard of care drugs for alcohol treatment and are not under study in this protocol.
  Computerized Brief Intervention (CBI): A video which emphasizes personal responsibility for change, uses empathy as a counseling style, and enhances self-efficacy. Depending on alcohol dependence level, four different CBI versions may be shown over two visits.
  CBT4CBT: 9 computerized modules delivered at the participant's pace Recommendation and Counseling for Alcohol Pharmacotherapy: The APT algorithm will utilize the four FDA approved APTs for the treatment of alcohol use disorder. The treatment of the patient is part of routine care.
Arm/Group | Risky Drinking, no dx of AUD, Has Panic or Depression | Dx of AUD With or Without Panic or Depression | No dx of Alcohol Use Disorder, Panic or Depression
Number analyzed (Participants) | 115 | 27 | 4843
score on a scale | -1.0 [-1.3 to -0.6] | -2.3 [-3.5 to -1.0] | -1.0 [-1.4 to -0.5]

2. Secondary Outcome: PEth Levels
Description: PEth is a biomarker for recent alcohol use found in the blood that is specific to ethanol ingestion and can detect low-to heavy drinking levels.
Time Frame: Between baseline and 6 month follow-up
Population: As a result of the COVID pandemic, sample collection was disrupted, leading to only 13 samples collected overall. This number of samples was below the 75% threshold needed to justify processing the samples. Samples were never sent for PeTH testing and will not be sent for PeTH testing.
Groups:
- No dx of Alcohol Use Disorder, Panic or Depre: Computerized Brief Intervention (CBI)- a video about alcohol abuse
  Computerized Brief Intervention (CBI): A video which emphasizes personal responsibility for change, uses empathy as a counseling style, and enhances self-efficacy. Depending on alcohol dependence level, four different CBI versions may be shown over two visits.
Arm/Group | No dx of Alcohol Use Disorder, Panic or Depre | Risky Drinking, no dx of AUD, Has Panic or Depression | Dx of AUD With or Without Panic or Depression
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 18 months
Arm/Group | Risky Drinking, no dx of AUD, Has Panic or Depression | Dx of AUD With or Without Panic or Depression | No dx of Alcohol Use Disorder, Panic or Depression
All-Cause Mortality (participants affected / at risk) | 0/115 | 0/27 | 0/4843
Serious Adverse Events (participants affected / at risk) | 0/115 | 0/27 | 0/4843
Other Adverse Events (participants affected / at risk) | 0/115 | 0/27 | 0/4843

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-23): https://cdn.clinicaltrials.gov/large-docs/77/NCT02938377/Prot_004.pdf
  • Informed Consent Form (2019-07-02): https://cdn.clinicaltrials.gov/large-docs/77/NCT02938377/ICF_002.pdf